CLINICAL TRIAL: NCT00556036
Title: Hormone Dynamics and Bone Mineral Density in Anorexia Nervosa v. Hypothalamic Amenorrhea
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Bioenvision (Industry)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital
Other Study IDs: 2003p-000549
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Anorexia Nervosa; Hypothalamic Amenorrhea; Obesity
Keywords: healthy; overweight; obese; anorexia nervosa; weight; cortisol; hormone; bone density; bone; osteopenia; osteoporosis; amenorrhea; menses; irregular; stress; depression; exercise; diet
MeSH Terms: conditions — Anorexia Nervosa; Obesity; Overweight; Body Weight; Bone Diseases, Metabolic; Osteoporosis; Amenorrhea; Depression; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood, serum, urine, saliva, optional DNA substudy.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: lean healthy women, age 18-45
- 2: overweight healthy women, age 18-45
- 3: women with hypothalamic amenorrhea (have not had a period in three months), age 18-45
- 4: women with anorexia nervosa, age 18-45

SUMMARY:
The purpose of this study is to determine whether the hormone dynamics in women with anorexia nervosa and hypothalamic amenorrhea is related to bone loss in those populations.

ELIGIBILITY:
Inclusion Criteria:

* Amenorrhea for at least three months (unless participating as healthy control)
* Normal TSH or free thyroxine (free T4).

Exclusion Criteria:

* A condition known to affect bone metabolism, including Cushing's syndrome or renal failure, with the exception of bone fracture.
* Any medication known to affect bone metabolism within 3 months of the study, including estrogen and progestins. Patients receiving depot medroxyprogesterone (Depo-Provera) will be excluded from participating for 6 months after their last injection.
* Pregnant and/or breastfeeding.
* Diabetes mellitus.
* Active substance abuse, including alcohol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample and referrals by specialists
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne A Klibanski, MD, Principal Investigator — Massachusetts General Hospital; Karen K Miller, MD, Study Director — Massachusetts General Hospital; Erinne M Meenaghan, NP, Study Chair — Massachusetts General Hospital; Elizabeth A Lawson, MD, Study Director — Massachusetts General Hospital; David B Herzog, MD, Study Chair — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States